CLINICAL TRIAL: NCT01966588
Title: Genomic Biomarkers of Adverse Events Arising From Antipsychotic Drug Therapy
Brief Title: Adverse Events and Genomics in Schizophrenia
Acronym: AEGIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health (Other Government); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: H13-00513
Record Dates: First submitted 2013-06-28; First posted 2013-10-21 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Adverse Effect of Other Antipsychotics and Neuroleptics
Keywords: Antipsychotic agents; Adverse effects; Genomics; Transcriptome
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — We will be collecting and retaining whole blood samples for genomic testing.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Metabolic Arm: Blood samples for whole genomic/transcriptomic sequencing; administration of the UKU Side Effect Rating Scale.
  Interventions: Other: Blood samples for whole genomic/transcriptomic sequencing; Other: UKU Side Effect Rating Scale
- Neutropenia/Immune System Arm: Blood samples for whole genomic/transcriptomic sequencing
  Interventions: Other: Blood samples for whole genomic/transcriptomic sequencing

INTERVENTIONS:
Other: Blood samples for whole genomic/transcriptomic sequencing — Participants in the Metabolic Arm will receive one blood draw, while participants in the Neutropenia Arm will receive a total of three blood draws: one at baseline, another 3 months later, and one 1 year later, with the possibility of further follow-up.
Other: UKU Side Effect Rating Scale — Clinician-rated scale of psychic, neurological, autonomic, and other side effects related to psychotropic drugs; ratings are based on a 10-30 minute interview with each participant.
  Other Names: UKU; Udvalg for Kliniske Undersøgelser
  Groups: Metabolic Arm

SUMMARY:
The purpose of this study is to find genes that predict whether or not a person will develop side effects to antipsychotic medications, such as weight gain, blood sugar dysregulation, or immune cell abnormalities. We will be collecting blood samples from participants who are taking second-generation antipsychotic medications. These blood samples will be stored over the long-term in a biobank, and will be used for later genetic testing and other cell-based studies.

DETAILED DESCRIPTION:
All data (including blood samples and medical information gathered from participants) will be labelled with each participant's unique coded identifier. Participants' identities will be matched with their coded identifier in a single, hard-copy of a Master Coding List. The maintenance and security of this list is the responsibility of the Principal Investigator.

All processing steps of the blood samples, including details of the blood draw, nucleic acid extraction, sequence library preparation, and sequence analysis will be documented in a Microsoft Excel worksheet. This worksheet will be encrypted for privacy.

Anonymized aliquots of blood samples (as well as any derived cell cultures) will be barcoded before long-term storage in a surveillance-monitored, secured freezer at -80 degrees Celsius. Samples within the freezer will be maintained via a positional numbered grid within the Laboratory Information Management System. This grid will also allow the study team to link each barcoded sample to a participant's coded identifier.

Mapped genomic sequences and other data collected from participants will be saved in password-protected folders on the UBC server. The coded sequence data will be transferred to the Department of Genetics and Genomic Sciences at Mount Sinai School of Medicine (MSSM) for further analyses. Data transfer will occur by Two Factor Identification. The MSSM secure network is Clinical Laboratory Improvement Amendments (CLIA) certified for secure handling of patient sequence data. The transfer of sequence data between UBC and MSSM will be performed under a material transfer agreement which requires that 1) all data and analysis be confined within the secure, password-protected database defined by UBC, 2) not distributed to any third party, and 3) both raw and analyzed data be destroyed from the MSSM monthly. This study is not required to comply with any U.S. federal regulations, as the group in MSSM will not have access to any identifying information about our participants.

ELIGIBILITY:
Inclusion Criteria:

* Must be taking an antipsychotic medication (no limit on treatment duration)

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals taking antipsychotic medications (in- or outpatients)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-06; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Concentration of whole-genome and/or transcriptome variants predicting weight gain, or glucose or lipid dysregulations in whole blood (ng/uL). | Anytime during a participant's course of treatment with second-generation antipsychotics (expected average of approximately 1 year after starting treatments)

SECONDARY OUTCOMES:
Concentration of whole-genome and/or transcriptome variants predicting immune effects of clozapine monotherapy in whole blood (ng/uL). | Baseline (at time of enrolment; expected average of approximately 1 year after starting treatment), 3 months after baseline, and 1 year after baseline (with possibility of further follow-up)

OTHER OUTCOMES:
Number of adverse effects, as rated by the UKU Side Effect Rating Scale. | Performed at the baseline blood draw for participants in both arms (at the time of enrolment into study; expected average of approximately 1 year after starting treatments)
  Adverse effects captured by the UKU include psychic/neurological/autonomic/and other side effects.
Frequency of side effects over the last 3 days, as measured by the UKU Side Effects Rating Scale | Performed at the baseline blood draw for participants in both arms (at the time of enrolment; expected average of approximately 1 year after starting treatments)

CONTACTS AND LOCATIONS:
Overall Officials: Alasdair M Barr, Ph.D., Principal Investigator — The University of British Columbia
Locations (1):
- BC Mental Health and Addictions Research Institute, Vancouver, British Columbia, Canada